CLINICAL TRIAL: NCT00000447
Title: Behavioral/Pharmacological Treatments for Alcohol-Nicotine Dependence
Brief Title: Behavioral/Drug Therapy for Alcohol-Nicotine Dependence (Naltrexone/Nicotine Patch)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: NIAAA-SCHMITZ-11216-04; R01AA011216 (NIH); NIH Grant 5R01AA011216-04
Record Dates: First submitted 1999-11-02; First posted 1999-11-03 (Estimated); Last update posted 2010-10-01 (Estimated); Status verified 2010-09

CONDITIONS: Alcoholism; Smoking
MeSH Terms: conditions — Alcoholism; Smoking | interventions — Naltrexone; Tobacco Use Cessation Devices

INTERVENTIONS:
Drug: naltrexone (Revia)
Drug: nicotine replacement patch

SUMMARY:
This study will develop a behavioral and drug relapse prevention program for individuals who are dependent on both alcohol and tobacco. The study's goal is to show that individuals receiving nicotine replacement therapy and naltrexone (Revia) with behavior therapy will have higher rates of abstinence from both smoking and drinking than individuals who do not receive the drug therapies. Individuals will be placed in a 12-week outpatient treatment program with followup assessments 1, 3, and 6 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for alcohol and nicotine dependence.
* Individuals will be outpatients with alcohol and nicotine dependence who have completed detoxification (medicated or nonmedicated) within the past 48-120 hours.
* Smoking no less than 10 cigarettes/day and no greater than 50 cigarettes/day.
* Motivated to quit smoking.
* Willing and able to participate in the 12 week outpatient treatment.
* Acceptable health.
* Able to provide a collateral informant.
* Willing to be followed for 6 months after treatment ends.
* Willing and able to provide the names of three family members or friends to aid in locating participants for follow-up.

Exclusion Criteria:

* Current diagnosis of dependence on other substances except nicotine and alcohol.
* Having moderately severe or severe alcohol withdrawal symptoms.
* Recent (less than 48 hours) evidence of hazardous drinking (more than 2 drinks/day for females; 3 drinks/day for males).
* History of opioid abuse.
* Recent use of cocaine.
* Not desiring to quit smoking.
* Recent past or current pharmacotherapy involving naltrexone or transdermal nicotine systems.
* History of psychosis.
* Current suicidality, homicidally or psychiatric symptoms requiring other medications.
* Presence of medical abnormalities that contraindicate naltrexone or nicotine replacement therapy.
* Current treatment with psychotropic medications.
* Pregnancy or nursing for female patients. Inability or unwillingness to participate in the 12-week outpatient treatment.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200
Dates: Start 1998-09; Study Completion 2003-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joy Schmitz, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Department of Psychiatry and Behavioral Sciences, University of Texas Health Science Center, Houston, Texas, United States